CLINICAL TRIAL: NCT03219450
Title: A Pilot Study of a Personalized Neoantigen Cancer Vaccine With and Without Low-Dose Cyclophosphamide or Pembrolizumab in Treatment Naïve, Asymptomatic Patients With IGHV Unmutated Chronic Lymphocytic Leukemia.
Brief Title: A Personalized Neoantigen Cancer Vaccine in Treatment Naïve, Asymptomatic Patients With IGHV Unmutated CLL.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Oncovir, Inc. (Industry); BioNTech SE (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Inhye Ahn, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 17-105
Record Dates: First submitted 2017-07-06; First posted 2017-07-17 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Lymphocytic Leukemia
Keywords: Leukemia; Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphoid; Leukemia | interventions — Cyclophosphamide; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- NeoVax (Experimental): * NeoVax will be administered in a priming and booster phase.
  * The priming shots will comprise days 1, 4, 8, 15, and 22.
  * Booster shots will be given on days 78 and 134.
  Interventions: Drug: NeoVax
- Neovax + Low-dose cyclophosphamide (Experimental): * NeoVax will be administered in a priming and booster phase.
  * The priming shots will comprise days 1, 4, 8, 15, and 22.
  * Booster shots will be given on days 78 and 134.
  * Low dose cyclophosphamide is administered twice daily on weeks -2, 1, 3, 5
  Interventions: Drug: NeoVax; Drug: Cyclophosphamide
- Neovax + Low-dose cyclophosphamide + Pembrolizumab (Experimental): * NeoVax will be administered in a priming and booster phase.
  * The priming shots will comprise days 1, 4, 8, 15, and 22.
  * Booster shots will be given on days 78 and 134.
  * Low dose cyclophosphamide is administered twice daily on weeks -2, 1, 3, 5
  * Pembrolizumab will be administered starting on Week 12 Day 78 and for up to 17 cycles (approximately 1 year).
  Interventions: Drug: NeoVax; Drug: Cyclophosphamide; Drug: Pembrolizumab

INTERVENTIONS:
Drug: NeoVax — It stimulates the immune system to attack cancer cells.
  Other Names: Neoantigen vaccine
Drug: Cyclophosphamide — It is a chemotherapy drug used to treat many cancers. At low doses, it is an investigational drug to help the immune cells to be better at attacking cancer cells while avoiding chemotherapy toxicity.
  Other Names: Cytoxan
  Arms: Neovax + Low-dose cyclophosphamide; Neovax + Low-dose cyclophosphamide + Pembrolizumab
Drug: Pembrolizumab — Is a monoclonal antibody that helps the immune cells to be better at attacking cancer cells.
  Other Names: Keytruda
  Arms: Neovax + Low-dose cyclophosphamide + Pembrolizumab

SUMMARY:
This research study is studying a novel type of CLL vaccine as a possible treatment for chronic lymphocytic leukemia (CLL)

The names of the study interventions involved in this study are:

* Personalized NeoAntigen Vaccine
* Poly-ICLC
* Cyclophosphamide
* Pembrolizumab

DETAILED DESCRIPTION:
This research study evaluates the feasibility and tolerability of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies. "Investigational" means that the intervention is being studied and that research doctors are trying to find more about it. It also means that the FDA (US Food and Drug Administration) has not approved the Personalized Neoantigen Cancer Vaccine for any use in patients, including people with CLL.

This is the first time NeoVax vaccine will be given in combination with cyclophosphamide and Pembrolizumab in humans.

The purpose of this study is to determine if it is possible to make and safely administer a vaccine against CLL. The investigators plan to analyze the specific genetic characteristics (mutations) of the participant's own CLL and use that information to produce proteins that may help the immune system recognize and fight CLL cells.

This vaccine is also being tested in clinical trials in patients with advanced melanoma (a type of skin cancer) or glioblastoma (a type of brain cancer). The current study will examine the ability of the vaccine to stimulate the immune system when given at several different timepoints, and will examine the participant blood cells for signs that the CLL has changed or decreased.

CLL cells will be obtained from bone marrow biopsy and blood draws. The genetic material contained in the CLL cells will be examined for the presence of tumor-specific mutations. This information will be used to prepare small protein fragments, which are called "peptides." The vaccine will consist of up to 20 of these peptides as well as a drug called Poly-ICLC. A peptide from the tetanus vaccine may also be included to boost the immune response. A third of the patients enrolled in this trial will receive the personalized neoantigen vaccine. Another third of the patients will also receive low doses of a chemotherapy drug called cyclophosphamide in combination of personalized neoantigen vaccine. The last third of patients enrolled in this study will receive the personalized neoantigen vaccine in combination with low dose cyclophosphamide and a drug called Pembrolizumab.

Poly-ICLC (also called Hiltonol) is an experimental "viral mimic" and an activator of immunity. Poly-ICLC binds proteins on the surface of certain immune cells to make it appear as if a virus is present. When the cells detect the vaccine, they think it is a virus and turn on the immune system. Poly-ICLC will be mixed with NeoAntigen peptides and administered as an injection given underneath the skin. Poly-ICLC is an investigational drug, meaning the FDA has not approved it as a treatment for any disease.

Cyclophosphamide (also called Cytoxan) is a chemotherapy drug used to treat many cancers, including CLL. At the much lower dose used in this study, it is an investigational drug to help the immune cells to be better at attacking cancer cells.

Pembrolizumab is a monoclonal antibody used to treat other types of cancer and information from these studies suggests that it may be beneficial in CLL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL as per IWCLL 2018 criteria
* Patient's CLL must have an unmutated immunoglobulin heavy chain variable (IGHV) region gene, defined as < 2% mutated compared to germline.
* Patient must have had no history of CLL-directed therapy due to meeting IWCLL 2018 criteria; no present indication for treatment by iwCLL 2018 criteria; and in the opinion of the treating investigator be anticipated not to require CLL-directed treatment within the next 6 months.
* Patient must have measurable disease (absolute lymphocyte count > 10K/uL or total white blood cell count ≥ 20K/uL of peripheral blood).
* Patient must have had at least two other absolute lymphocyte counts (ALC) measured since diagnosis of CLL that are at least 2 weeks apart and at least 2 months prior to the one used for initial registration.
* Age ≥ 18 years.
* ECOG performance status 0 or 1
* Participants must have normal organ and marrow function as defined below:

  * total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
  * absolute neutrophil count ≥1000 cells/μL
* The effects of NeoVax and poly-ICLC on the developing human fetus are unknown. For this reason, women of childbearing potential (WOCBP) must have a negative pregnancy test (minimum sensitivity 25 IU/L or equivalent of HCG) before entry onto the trial and within 7 days prior to start of study medication. It is the investigators' responsibility to repeat the pregnancy test should start of treatment be delayed.
* Female patients enrolled in the study, who are not free from menses for >2 years, post hysterectomy / oophorectomy, or surgically sterilized, must be willing to use either 2 adequate barrier methods or a barrier method plus a hormonal method of contraception to prevent pregnancy or to abstain from sexual activity throughout the study, starting with visit 1 through 4 weeks after the last dose of study therapy. Approved contraceptive methods include for example; intra uterine device, diaphragm with spermicide, cervical cap with spermicide, male condoms, or female condom with spermicide. Spermicides alone are not an acceptable method of contraception.
* Patient is agreeable to allow tumor (from peripheral blood) and normal tissue (from saliva) samples to be submitted for complete exome and transcriptome sequencing.
* Ability to understand and the willingness to sign a written informed consent document.
* At least 7 immunizing peptides can be designed.
* Continue to meet inclusion and exclusion criteria for Screening Registration.

Exclusion Criteria:

* Prior therapy for CLL that met IW-CLL treatment criteria, including chemotherapy, targeted therapies (e.g. that antagonize B cell receptor signaling), or immunotherapy (including but not limited to monoclonal antibodies); or radiotherapy or hormonal therapy within the last 2 years of screening registration.
* Participants who are receiving any other investigational agents.
* Previous bone marrow or stem cell transplant
* Concomitant therapy with immunosuppressive or immunomodulatory agents; chronic use of systemic corticosteroids. Previous history of corticosteroid use is acceptable. Use of corticosteroids after initial registration is acceptable if tapered at least one week before NeoVax administration.
* Use of a non-oncology vaccine therapy for prevention of infectious diseases within 2 weeks of any NeoVax administration.
* History of severe allergic reactions attributed to any vaccine therapy for the prevention of infectious diseases.
* Participants who have never received the tetanus vaccine.
* Active, known, or suspected autoimmune disease or immunosuppressive conditions with the exception of vitiligo, type 1 diabetes, residual autoimmune-related hypothyroidism requiring hormone replacement, or psoriasis not requiring systemic treatment.
* Uncontrolled autoimmune cytopenia.
* No lymph node > 5 cm by CT scan (measured as long axis).
* Del(17p) by fluorescence in situ hybridization in ≥ 10% of CLL cells analyzed
* Any documented transformation of CLL (i.e. Richter's Syndrome).
* Lymphocyte doubling time (LDT) < 6 months in patients with WBC > 30,000/uL. Factors contributing to lymphocytosis other than CLL (e.g. infections) should be excluded when calculating the LDT1.
* Serum immunoglobulin level <400 mg/dL or currently requiring chronic intravenous immunoglobulin G (IVIG)
* Known chronic infections with HIV, hepatitis B or C (see Study Calendar in Section 10 for screening assays).
* Has received prior therapy with an anti-PD1, anti PD-L1, or anti PD-L2 agent.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia.
* Any underlying medical condition, psychiatric condition or social situation that in the opinion of the investigator would compromise study administration as per protocol or compromise the assessment of AEs.
* Pregnant women are excluded from this study because personalized neoantigen peptides and poly-ICLC are agents with unknown risks to the developing fetus. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with personalized neoantigen peptides and poly-ICLC, nursing women are excluded from this study.
* Individuals with history of an invasive malignancy are ineligible except for the following circumstances: a) individuals with a history of invasive malignancy are eligible if they have been disease -free for at least 3 years and are deemed by the investigator to be at low risk for recurrence of that malignancy; b) individuals with the following cancers are eligible if diagnosed and treated: carcinoma in situ of the breast, oral cavity or cervix and basal cell or squamous cell carcinoma of the skin; c) individuals with prostate cancer managed with active surveillance that is not expected to limit their survival to <10 years.
* Participants with known CNS involvement should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to poly-ICLC.
* HIV-positive participants on combination antiretroviral therapy are ineligible because assessment of immunologic endpoints may be confounded by HIV-induced alterations in patient immune status and function. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-08-18 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of neoantigen identification | 6 months
  The proportion of all enrolled patients for whom sequencing and analysis leads to identification of at least 7 actionable peptides to initiate vaccine production
Feasibility of vaccine generation | 6 months
  Of the patients who generate at least 7 actionable peptides, the proportion for whom the time from sample collection to vaccine availability is less than 12 weeks
Safety of NeoVax | 1 year
  The number of patients with treatment-limiting toxicities based on NCI CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Inhye Ahn, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No